CLINICAL TRIAL: NCT04937309
Title: Efficacy and Safety of Non Invasive Vagal Stimulation to Prevent Chemotherapy-induced Nausea in Patients With Breast Cancer Receiving Anthracycline and Cyclophosphamide Chemotherapy
Brief Title: Efficacy and Safety of Non Invasive Vagal Stimulation to Prevent Chemotherapy-induced Nausea
Acronym: SILENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DR210090_SILENCE
Record Dates: First submitted 2021-06-03; First posted 2021-06-24 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: nausea; non invasive vagal stimulation; chemotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Nausea

STUDY DESIGN:
Intervention Model Description: one control arm and one intervention arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sham
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): standard anti emetic treatment use of non invasive vagal stimulation twice a day from the day before chemotherapy till 4 days after, with a transcutaneous auricular device. This stimulation is to be done for the three first cycles of chemotherapy.
  Interventions: Device: non invasive auricular vagal stimulation; Drug: usual medical treatment
- control (Sham Comparator): standard anti emetic treatment use of non invasive vagal stimulation twice a day from the day before chemotherapy till 4 days after, with a transcutaneous auricular sham device. This "stimulation" is to be done for the three first cycles of chemotherapy.
  Interventions: Drug: usual medical treatment; Device: sham stimulation

INTERVENTIONS:
Device: non invasive auricular vagal stimulation — Stimulation twice a day, beginning the day before until the fourth day after chemotherapy, for the three first chemotherapy cycles
  Arms: intervention
Drug: usual medical treatment — Standard anti emetic treatments to prevent emesis due to chemotherapy
Device: sham stimulation — Stimulation twice a day, beginning the day before until the fourth day after chemotherapy, for the three first chemotherapy cycles, with a sham device
  Arms: control

SUMMARY:
Despite pharmaceutical innovations, chemotherapy induced nausea is frequent and largely participating to alter our patients quality of life.

Non invasive vagal stimulation is approved in other health issues, for example in headache or gastroparesis, with a reported benefit on nausea.

This study aims to analyse if a non invasive vagal stimulation could better prevent chemotherapy induced nausea, in addition to standard treatment, in breast cancer patients treated with cyclophosphamide and anthracycline.

DETAILED DESCRIPTION:
Despite pharmaceutical innovations, chemotherapy induced nausea is frequent and largely participating to alter our patients quality of life.

Non invasive vagal stimulation is approved in other health issues, for example in headache or gastroparesis, with a reported benefit on nausea.

This study aims to analyse if a non invasive vagal stimulation could better prevent chemotherapy induced nausea, in addition to standard treatment, in breast cancer patients treated with cyclophosphamide and anthracycline.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) status 0 to 2
* patient with breast cancer planned to receive Anthracycline and Cyclophosphamide chemotherapy
* informed consent
* compliance expected
* social security affiliation

Exclusion Criteria:

* nausea or vomiting 24h or less, before inclusion
* Antiemetic drug intake in the last 72h before inclusion
* Central nervous system metastasis
* Daily alcohol intake
* Prior chemotherapy
* Cardiac arrythmia, severe heart failure
* Device for sleep apnea
* History of arterial or venous thrombosis, or thrombophlebitis
* Vagotomy
* Vagal stimulation ongoing
* Skin disease on the stimulation zone
* Cochlear implant next to the stimulation zone
* Unable to use the vagal stimulation device due to left ear unusual shape
* Pregnant or breastfeeding women, or women of childbearing age without effective contraception
* Documented allergy or contraindication to one of the antiemesis drugs required in the study
* Protected adults (individuals under guardianship by court order)
* Unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with significant nausea after the first chemotherapy cycle | 2 to 3 weeks
  Nausea severity is graded daily from Day 1 (day of chemotherapy) to Day 5, using a numeric scale from 0 to 10. It is a patient reported outcome, patients using a diary. Significant nausea is a score of 2 or more.

SECONDARY OUTCOMES:
Percentage of patients with significant nausea after the second and the third chemotherapy cycle. | 7 to 12 weeks
  Same measurement at the second and the third chemotherapy. And global score considering the three cycles together.
Percentage of patients that did not vomit or use rescue emesis medication, from the first cycle of chemotherapy to day 5 after the third chemotherapy cycle. | 7 to 12 weeks
  Percentage of patients without any vomiting, or rescue emesis medication use, from first to third chemotherapy
Percentage of non planned visit to emergency care unit or general practioner or oncologist due to emesis, measured for the three first chemotherapy cycles. | 7 to 12 weeks
  To measure complication due to emesis from the first cycle of chemotherapy to day 5 after the third chemotherapy cycle
Percentage of non anticipated hydratation with IV fluids measured for the three first chemotherapy cycles. | 7 to 12 weeks
  To measure complication due to emesis from the first cycle of chemotherapy to day 5 after the third chemotherapy cycle
Percentage of hospitalisations for emesis measured for the three first chemotherapy cycles. | 7 to 12 weeks
  To measure complication due to emesis from the first cycle of chemotherapy to day 5 after the third chemotherapy cycle
quality of life measurement using international validated questionnaire EORTC QLQ-C30 (quality of life questionnaire -C30), EORTC QLQ-BR23 (quality of life questionnaire for breast cancer), completed at the first three cycles | 9 to 15 weeks
  patient reported outcome measure, using international validated questionnaires and patient diaries
number and type of side effect during vagal stimulation safety | 7 to 12 weeks
  report of any side effect, based on patient declaration

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CH BLOIS, Blois
  - Chru Morvan, Brest
  - CORT37, Chambray-lès-Tours
  - Ch Chateauroux, Châteauroux
  - Clinique Victor Hugo, Le Mans
  - Ch Orleans, Orléans
  - Ch Chinon, Saint-Benoît-la-Forêt
  - CHRU Bretonneau, Tours